CLINICAL TRIAL: NCT01795144
Title: Incretin Regulation of Insulin Secretion in Monogenic Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 12-1517
Record Dates: First submitted 2013-02-15; First posted 2013-02-20 (Estimated); Last update posted 2017-04-10 (Actual); Status verified 2017-04

CONDITIONS: Monogenic Diabetes
MeSH Terms: interventions — Glucagon-Like Peptide 1; exendin (9-39)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healthy controls (Active Comparator): Healthy controls will be matched (age, gender, BMI) to monogenic diabetes subjects. Healthy controls will participate in the following:
  * OGTT
  * IGI
  * IGI with GLP-1 infusion
  * OGTT with Exendin 9-39 infusion
  Interventions: Drug: GLP-1; Drug: Exendin 9-39
- Monogenic diabetes (Experimental): Monogenic diabetes subjects will be matched (age, gender, BMI) to healthy controls. Monogenic diabetes subjects will participate in the following:
  * OGTT
  * IGI
  * IGI with GLP-1 infusion
  * OGTT with Exendin 9-39 infusion
  Interventions: Drug: GLP-1; Drug: Exendin 9-39

INTERVENTIONS:
Drug: GLP-1 — OGTT IGI IGI with GLP-1 infusion OGTT with Exendin 9-39 infusion
  Other Names: Glucagon-like peptide-1 (GLP-1)
Drug: Exendin 9-39 — OGTT IGI IGI with GLP-1 infusion OGTT with Exendin 9-39 infusion
  Other Names: Glucagon-Like Peptide 1 (GLP-1) receptor antagonist

SUMMARY:
The purpose of this study is to explore the mechanisms of metabolic control in monogenic diabetes patients treated with sulfonylurea medications.

DETAILED DESCRIPTION:
Monogenic diabetes patients and healthy matched controls will be admitted to the University of Chicago Clinical Resource Center for a total of 4 nights. The following will take place on separate days:

1. Oral Glucose Tolerance Test (OGTT): consume sugary drink and blood samples will be collected at multiple time points
2. Isoglycemic glucose infusion (IGI) test: glucose will be infused via a vein in the arm and and blood samples will be collected at multiple time points
3. OGTT during GLP-1 infusion
4. IGI during Exendin-9 infusion

ELIGIBILITY:
Monogenic Diabetes Subjects:

Inclusion Criteria:

* Diagnosis of monogenic diabetes
* Previously participated in US Neonatal Diabetes Registry (IRB 15617B) or Genetics of diabetes mellitus (IRB 6858)
* Age: 18 years +

Exclusion Criteria:

* Pregnancy
* Acute medical illness or chronic conditions including: cardiac failure, renal insufficiency (estimated glomerular filtration rate <50 ml/min), hepatic insufficiency (known cirrhosis or hepatitis), chronic obstructive pulmonary disease, gastrointestinal disorders causing malabsorption, anemia (Hct < 36%), or uncontrolled hypertension

Healthy Controls:

Inclusion Criteria:

* Good general health
* Stable weight for 6 months
* Age: 18 years +

Exclusion Criteria:

* Pregnancy
* Acute medical illness or chronic conditions including: cardiac failure, renal insufficiency (estimated glomerular filtration rate <50 ml/min), hepatic insufficiency (known cirrhosis or hepatitis), chronic obstructive pulmonary disease, gastrointestinal disorders causing malabsorption, anemia (Hct < 36%), or uncontrolled hypertension

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-01; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Incretin Effect | Baseline
  Directly calculated from the difference between oral and IV stimulated insulin secretion

CONTACTS AND LOCATIONS:
Overall Officials: Siri Atma W Greeley, MD, PhD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
We do not plan to share data with other researchers.